CLINICAL TRIAL: NCT03970642
Title: Video Directly Observed Therapy (VDOT) to Improve Medication Adherence Among Depression Patients
Brief Title: Video Directly Observed Therapy (VDOT) to Improve Medication Adherence
Acronym: NARSAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment closed early due to Covid-19.
Sponsor: UConn Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 19-136-2
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Depression
Keywords: video directly observed therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: In this randomized controlled trial, participants will be randomly assigned to the study or the control group. A total of up to 100 participants will be enrolled (50 participants assigned to each group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive individualized text reminders on their phone prior to each dose of their depression medicine. They will receive the video directly observed therapy smartphone app. Research staff will be able to monitor these medication adherence video on a password protected server linked to the app. Upto 50 patients will be randomly assigned to this group.
  Interventions: Other: Video directly observed therapy
- Control (No Intervention): The control group will receive current standard of care. Upto 50 patients will be randomly assigned to this group.

INTERVENTIONS:
Other: Video directly observed therapy — The intervention group will receive individualized text reminders on their phone prior to each dose of their depression medicine. They will be requested to use the VDOT smartphone app to make a video recording of each medication dose ingested during the 3 month study period following their first visit. The app will automatically upload the video to a HIPAA compliant server. Research staff will regularly monitor videos using a password protected website and document each medication dose.
  Arms: Intervention group

SUMMARY:
Due to the lack of human resources, it is impossible to monitor patients' medication adherence objectively or in-person by observation like tuberculosis programs worldwide do. The feasibility and patient acceptance of the innovative video-based directly observed therapy (VDOT) approach for improving medication adherence among tuberculosis patients has been demonstrated through studies in the United States as well as internationally (7). Medication adherence among VDOT users has been found to be comparable to in-person directly observed treatment (91% vs 95%) among patients in New York (8). In this clinical research project, we will test the feasibility, acceptance and effectiveness of an innovative mobile-based behavioral intervention to improve medication adherence and depression symptoms among patients suffering from depression.

DETAILED DESCRIPTION:
This is a randomized prospective study utilizing Video Directly Observed Therapy (VDOT), which is a novel means of remotely observing patients ingesting medications using videos sent from the patients' smartphone application. The VDOT mobile phone application called SureAdhere was developed and found to be feasible and acceptable for monitoring daily treatment of active tuberculosis in San Diego, CA (R21-AI088326; PI: R. Garfein). For testing the feasibility, acceptance and effectiveness of VDOT application (app) SureAdhere among depression patients, we will conduct a two-arm randomized controlled trial for which a maximum of 100 patients will be recruited (50 patients in study group; 50 patients in control group). Informed consent will be obtained prior to the start of study activities.Randomization will be performed using a computer generated randomization program assigning a random group to each consecutive study participant. This will be performed prior to the study and stored in a list with participant numbers. Those assigned to the control group will receive care as usual. Those assigned to study group will receive assistance in installing the SureAdhere app on their own smartphone. If they did not own a smartphone, a loaned smartphone with internet service plan and preinstalled SureAdhere mobile phone application will be provided to them if available. The SureAdhere app is programmed to send encrypted, time/date stamped videos to a HIPAA-compliant server. The study group subjects will receive a pin for their individualized log-in through a text message on their phone. They will be trained on how to use the application to send videos through a training video and handouts provided to them. Study staff will be available to answer any questions or concerns about the SureAdhere app. In case of technical issues, study staff will gather information about the concerns and then get input from the customer support team at SureAdhere, Inc. to resolve the issues. The study group subjects will receive individualized text reminders on their phone prior to each dose of their depression medicine. They will be requested to use the VDOT smartphone app to make a video recording of each medication dose ingested during the 3 month study period following their first visit. Research staff will regularly monitor videos using a password protected website and document each medication dose. Outcomes data will be obtained through self-report questionnaires at three time points: baseline, about 6 weeks and about 3 months and from the patient medical records. The baseline questionnaire will be conducted after the informed consent and will collect information about demographic characteristics (i.e. date of birth, sex, race, ethnicity, type of residence- house vs apartment own vs rent, type of insurance), medication adherence (using ASK-20 Medication Adherence questionnaire) and depression symptoms (using Patient Health Questionnaire-9). Both these validated survey tools are available for public use. The follow-up questionnaires sent to the subjects will obtain additional information regarding technology acceptance from the participants in the study group only. From all subjects, the follow-up questionnaires will gather information about medication adherence and depression symptoms. Patient medical records and VDOT video review will be used to obtain an objective measure of medication adherence, comorbidities (Elixhauser co-morbidity score) and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be English speaking
* >=18 years old
* diagnosed with depression and currently prescribed oral antidepressant medication
* own a mobile phone and active phone plan capable of receiving text messages.

Exclusion Criteria:

* Non-English speakers, minors (<18 years old)
* patients diagnosed with bipolar disorder (patient may be included if the study team determines that the historical diagnosis of bipolar disorder was inaccurate)
* visual or cognitive disabilities and/or terminal illness
* patients with any clinically significant medical or psychiatric condition, as deemed by the investigator, that can affect their ability to participate in the protocol, including primary psychotic disorder, and active suicidal intent or plan at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Change in medication adherence | The questionnaire will be administered at baseline, 6 weeks and 3 months.
  The change in medication adherence during the study period will be determined using the ASK-20 questionnaire. The ASK-20 questionnaire includes 20 questions, each with a likert response from 1 to 5 with 1 representing excellent and 5 representing poor medication adherence.

SECONDARY OUTCOMES:
Change in depression symptoms | The questionnaire will be administered at baseline, 6 weeks and 3 months.
  The PHQ9 questionnaire will be used to examine the change in depression symptoms. This 9-question scale has a four point likert scale with 1 being the least and 4 representing the highest depression symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- UConn Health Psychiatry practice, Farmington, Connecticut, United States